CLINICAL TRIAL: NCT01428674
Title: The Impact of Interpersonal Mindful Compassion on Autonomic Nervous System Function
Brief Title: Time, Touch, Attention and the Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00015699
Record Dates: First submitted 2011-08-30; First posted 2011-09-05 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Stress
Keywords: Interpersonal mindful compassion; Loving kindness meditation; Autonomic Nervous System; Heart rate variability; Respiratory rate; Relaxation
MeSH Terms: interventions — Touch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 10 minutes reading (Experimental)
  Interventions: Other: Reading while extending loving kindness
- 20 minutes touch (Experimental)
  Interventions: Other: Interpersonal Mindful Compassion with Touch
- 20 minutes reading (Experimental)
  Interventions: Other: Reading while extending loving kindness
- 10 minutes touch (Experimental)
  Interventions: Other: Interpersonal Mindful Compassion with Touch

INTERVENTIONS:
Other: Interpersonal Mindful Compassion with Touch — A practitioner lightly touches the participant on the hands, arms, shoulders, lower legs and feet while extending loving kindness to the participant.
  Arms: 10 minutes touch; 20 minutes touch
Other: Reading while extending loving kindness — The practitioner sits in a room with the participant, pretending to read, while extending loving kindness to the participant.
  Arms: 10 minutes reading; 20 minutes reading

SUMMARY:
The purpose of this study is to describe the onset, duration and dose-response of interpersonal mindful compassion on respiratory rate and heart rate variability in healthy adults in order to prepare for research evaluating the impact of this intervention in patient populations and to prepare for basic research investigating the CNS mechanisms for observed effects.

Previous research has found that mindfulness meditation, including mindful compassion, results in autonomic changes in the practitioner. Emerging neuroscience of dyadic interactions suggests that through the effects of mirror neuron isopraxis, one person's physiologic state may be mirrored by another. However, no research has directly evaluated the impact of one person's mindful compassion on another person's autonomic activity. This study paves the way for an entirely new avenue of research inquiry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects age 18 - 40

Exclusion Criteria:

* Taking beta blocker medication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate Variability from pre-intervention period to intervention period | continuous monitoring for 10 min before intervention and during 10 or 20 minute intervention
Change in Respiratory Rate from pre-intervention period to intervention period | continuous monitoring for 10 minutes before intervention and during 10 or 20 minute intervention

SECONDARY OUTCOMES:
Perceived Stress, Relaxation, Peacefulness | baseline, after a 10 minute rest period, before 10 or 20 minute intervention, immediately after intervention, 20 minutes after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kathi J Kemper, MD, Principal Investigator — Wake Forest University Health Sciences

REFERENCES:
- [Derived] Kemper KJ, Shaltout HA. Non-verbal communication of compassion: measuring psychophysiologic effects. BMC Complement Altern Med. 2011 Dec 20;11:132. doi: 10.1186/1472-6882-11-132. PMID 22185349